CLINICAL TRIAL: NCT06881186
Title: The Use of Collagen-based Filler for Trapeziometacarpal Osteoarthritis. Long-term Follow Up and Future Applications
Brief Title: Collagen-based Filler for Trapeziometacarpal Osteoarthritis
Status: Completed | Type: Observational
Sponsor: Azienda Ospedaliera Universitaria Integrata Verona (Other)
Responsible Party: Principal Investigator, Massimo Corain, Principal Investigator, Azienda Ospedaliera Universitaria Integrata Verona
Other Study IDs: 3185CESC
Record Dates: First submitted 2025-02-11; First posted 2025-03-18 (Actual); Last update posted 2025-03-18 (Actual); Status verified 2025-02

CONDITIONS: Trapeziometacarpal Osteoarthritis
MeSH Terms: interventions — Injections, Intra-Articular

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

INTERVENTIONS:
Procedure: Intra-articular injection — Intra-articular injection of a cell-free collagenic gel matrix into the trapeziometacarpal joint

SUMMARY:
Introduction. Trapeziometacarpal osteoarthritis (TMC OA) is a degenerative condition characterized by pain, stiffness, and reduced hand function, significantly impairing daily activities. Non-surgical management strategies include activity modifications, nonsteroidal anti-inflammatory drugs (NSAIDs), splinting, and corticosteroid injections. When conservative treatments fail, surgical options are considered. The Eaton-Littler classification stratifies TMC OA into four stages based on radiographic joint degeneration.

ChondroFiller Liquid®, a cell-free collagen scaffold composed of native type I collagen and chondrostimulating factors, facilitates cartilage regeneration by creating a protective environment for chondrocyte proliferation. It is indicated for treating cartilage lesions up to 3 cm². A prior study demonstrated its efficacy in alleviating pain, improving grip strength (Jamar test and pinch test), and enhancing Patient-Reported Outcome Measures (PROMs) using the Disabilities of the Arm, Shoulder, and Hand (DASH) score.

Aims. This study aims to extend the follow-up to 24 months to evaluate the long-term sustainability of clinical improvements following ChondroFiller Liquid® infiltration.

Materials and Methods. A total of 40 patients from the initial study were enrolled and categorized into two severity groups based on the Eaton-Littler classification. Clinical evaluations were conducted at 18 months post-infiltration (T1) using the Numeric Rating Scale (NRS) and DASH score. A subsequent assessment at 24 months (T2) included the Jamar test, pinch test, NRS, and DASH score. An additional cohort of 51 patients underwent infiltration with a mean follow-up of 14 months, including 9 patients previously treated in the preliminary study.

ELIGIBILITY:
Inclusion Criteria:

* patients with rhizarthrosis diagnosed on X-rays performed in the last year;
* patients aged > 18 years;
* enrollment in the study through informed consent;

Exclusion Criteria:

* patients who have undergone cortisone and/or hyaluronic acid infiltrations in the last 6 months;
* patients following trauma involving the ATM;
* patients with underlying rheumatological diseases;
* patients under 18 years of age
* ongoing pregnancy;
* patients affected by metabolic disorders (e.g. diabetes)

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All participants were adults with unilateral or bilateral RA, diagnosed via radiographs obtained within the past year. Participation in the study required signing an informed consent form.
Sampling Method: Non-Probability Sample
Enrollment: 64 (Actual)
Dates: Start 2021-01-01 (Actual); Primary Completion 2023-01-01 (Actual); Study Completion 2025-01-01 (Actual)

PRIMARY OUTCOMES:
DASH (Disabilities of the Arm, Shoulder, and Hand) | 2 years
  The DASH is a self-administered questionnaire of over 30 questions designed to measure function and symptoms in patients with any musculoskeletal disorder of the upper limb. MAX 100, MIN 0
VAS (Visual Analogue Scale) | 2 years
  The pain VAS is a unidimensional measure of pain intensity, used to record patients' pain progression, or compare pain severity between patients with similar conditions. MAX 10, MIN 0
Jamar test | 2 years
  The Jamar test consists of evaluating grip strength using a hand dynamometer. MIN 0 MAX 100 Kgm.
Pinch tests | 2 years
  The Pinch tests consist of three tests assessed with a specific dynamometer, evaluating the two-finger grip, three-finger grip, and key grip. MIN 0, MAX 15 Kgm.

CONTACTS AND LOCATIONS:
Locations (1):
- Azienda Ospedaliera Universitaria Integrata, Verona, ITA, Italy

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Corain M, Faccioli N, Lavagnolo U. The Use of Collagen-Based Filler for Trapeziometacarpal Osteoarthritis: Long-Term Follow-Up and Future Applications. Cartilage. 2025 Jul 1:19476035251354926. doi: 10.1177/19476035251354926. Online ahead of print. PMID 40590316